CLINICAL TRIAL: NCT06194097
Title: Management of Pediatric Chronic Rhinosinusitis in Asthmatic Children
Brief Title: Pediatric Chronic Rhinosinusitis in Asthmatic Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: poor recruitment
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1009628-5
Record Dates: First submitted 2017-11-01; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2021-04

CONDITIONS: Sinusitis in Children
MeSH Terms: interventions — Adenoidectomy

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adenoidectomy (Experimental)
  Interventions: Procedure: adenoidectomy versus endoscopic sinus surgery with adenoidectomy
- Endoscopic Sinus surgery and Adenoidectomy (Experimental)
  Interventions: Procedure: adenoidectomy versus endoscopic sinus surgery with adenoidectomy

INTERVENTIONS:
Procedure: adenoidectomy versus endoscopic sinus surgery with adenoidectomy — adenoidectomy versus endoscopic sinus surgery

SUMMARY:
The objectives of this study would be to determine the most effective treatment for children with PCRS and asthma who fail medical management.

DETAILED DESCRIPTION:
This prospective, randomized study would involve children age 6-12 with symptoms of both PCRS and asthma. Their symptoms would first be managed medically with standard medical therapy. In the event they fail medical management, patients would then be randomized to two treatment arms, either adenoidectomy alone or adenoidectomy with ESS. CT scan of the sinuses would then be obtained to evaluate the extent of sinus disease and aid in preoperative planning in those patients undergoing ESS. Sinus mucosa thickening seen on CT is also integral in the diagnosis of PCRS, according to consensus statements published by the American Academy of Otolaryngology. At each visit patient's symptoms would be measured with the SN-5, a validated questionnaire for tracking PCRS.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

Age 6-12 at time of study enrollment. Presence of chronic sinusitis: >90 days 2 or more symptoms of purulent rhinorrhea, nasal obstruction, facial pressure/pain, or cough with corresponding endoscopic and/or CT findings in a patient 18 years or younger.

Presence of asthma, as documented in the medical record by the patient's pediatrician and/or pulmonologist

Exclusion Criteria:

* Exclusion criteria include previous sinus surgery, previous adenoidectomy, or presence of cystic fibrosis, antrochoanal polyp, immunodeficiency, or fungal infection.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2020-07-25 (Actual); Study Completion 2020-07-25 (Actual)

PRIMARY OUTCOMES:
surgical outcome | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY Upstate Medical Center, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No